CLINICAL TRIAL: NCT02628314
Title: Reliability of Pupil Response to Acute Pain
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00033891
Record Dates: First submitted 2015-07-08; First posted 2015-12-11 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pain; Osteoarthritis
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osteoarthritis: Study population to include adult men and women with osteoarthritis.

SUMMARY:
The purpose of this research study is to test whether researchers can reliably measure the response pupils have when an acute painful stimulus is experienced. Changes in the size of the pupil of the eye can be an indicator of brain activity in a region of the brain that is important for feeling pain.

DETAILED DESCRIPTION:
There is strong rationale to support a role for locus coeruleus (LC) responsivity to acute painful stimuli in regulating speed of recovery after surgery and for LC responsivity as a mechanistic link explaining the risks for slow recovery from weak Conditioned Pain Modulation (CPM), catastrophizing cognitive style, and low enzyme activity catecholamine-O-methyltransferase (COMT) genotype. Preliminary data show feasibility to perform the proposed study.

Primary Hypothesis: An observational study of pupil responses to noxious stimuli shows strong intra-individual reliability over 8 weeks.

Key secondary hypotheses: Compared to individuals homozygous for val at the val158met site of the catecholamine-O-methyltransferase (COMT) gene, those homozygous for met will show smaller pupil responses to noxious stimuli and weaker CPM.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-70)
* Pain from hip or knee arthritis of moderate intensity
* American Society of Anesthesiologists physical status 1-3

Exclusion Criteria:

* Inability to complete study questionnaires
* Pregnancy
* Litigation or workers compensation related to hip or knee pain
* Taking > 50 mg morphine equivalents/day
* History of Raynaud's disease of the feet
* Psychotic disorder or a recent psychiatric hospitalization
* History of eye surgery or topical eye medications that would would directly affect pupil diameter

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with athritis in the knee or hip with moderate average daily pain score
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-08-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of change in pupil diameter | 8 weeks
  pupil diameter in response to 5 second presentation of noxious heat stimuli
Change from Baseline Verbal Pain Scores | 8 weeks
  Verbal pain scores will be obtained during stimulus presentation

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States